CLINICAL TRIAL: NCT06296550
Title: Enhancing Digitally Delivered Diabetes Education With Real-Time CGM: A Comparative Study in People With Type 2 Diabetes
Brief Title: Enhancing Digitally Delivered Diabetes Education With Real-Time CGM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Whittier Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dulce Digital CGM
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Type 2
Keywords: Diabetes; CGM; Diabetes Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGM Group (Experimental): Participants will be provided continuous glucose monitors (Dexcom G7) to monitor blood glucose for the entire duration of this study (i.e., one new device every 10 days for a total of 18 devices to last up to 6 months).
  Interventions: Other: Dulce Digital Text Messaging Intervention; Other: CGM Device
- Usual Care Blood Glucose Monitoring Group (Other): Participants will use standard blood glucose monitoring devices that are covered by health insurance.
  Interventions: Other: Dulce Digital Text Messaging Intervention

INTERVENTIONS:
Other: Dulce Digital Text Messaging Intervention — Text-based education support program:
  * Participants will receive text messages about diabetes and how to take care of diabetes and health. Participants will receive 2-3 messages every day for first 3 months, and then will slowly decrease over the last 3-months.
  * Participants will also receive text messages that will ask them to test their blood sugar and text back blood sugar reading.
Other: CGM Device — Participants will be provided continuous glucose monitors (Dexcom G7) to actively monitor blood glucose for the entire duration of this study (i.e., one new device every 10 days for a total of 18 devices to last up to 6 months). In addition, participants will attend an information session (group or individual; in-person or virtual) that will provide instructions on using continuous glucose monitors.
  Arms: CGM Group

SUMMARY:
The current research study will add continuous glucose monitoring devices to the evidence-based text messaging diabetes education program for patients with type 2 diabetes for 6 months. Results on the effectiveness of this intervention will be compared for non-insulin using patients.

DETAILED DESCRIPTION:
The current research study seeks to investigate the impact of incorporating Continuous Glucose Monitoring (CGM) into the evidence-based text messaging diabetes education program, Dulce Digital, focusing on individuals with Type 2 Diabetes (T2D) who are not on insulin therapy. This innovative approach stems from the rationale that real-time continuous glucose monitoring (CGM) can offer valuable insights into glycemic control, thereby enhancing diabetes self-management. In standard care, individuals with T2D, particularly those not on insulin, may not routinely have access to CGM devices. The CGM device, an integral part of recommended diabetes therapy, is FDA approved for use in all people with diabetes. However, reimbursement for CGM devices varies by health plans, and currently, Centers for Medicare & Medicaid Services (CMS) does not reimburse for their use in non-insulin-using diabetes, except in cases of repeated severe hypoglycemia. Despite this, the investigators hypothesize that there are both clinical and financial benefits to providing a CGM device during diabetes self-management education for individuals with non-insulin-using T2D. This study aims to determine if adding a CGM device for this patient category yields significant benefits, contributing to the understanding of the potential advantages and informing future diabetes care practices.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Are not currently using a CGM
* Are not using insulin therapies
* Speak English, Spanish or Arabic
* Have A1c between 7.5% and 12.0% in last 90 days
* Have a cellphone that can receive/send text messages and counts steps

Exclusion Criteria:

* Are using insulin therapies
* Are pregnant
* Are currently using a CGM
* Are currently participating in another diabetes-related study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 6 months
  Measures participants A1c using lab results provided from healthcare provider.

SECONDARY OUTCOMES:
CGM Metric Time in Range | 6 months
  Measures the percentage of time a participant's blood glucose levels stay within the target range using CGM device.
CGM Metric Time above Range | 6 months
  Measures the percentage of time a participant's blood glucose levels exceed the target range using CGM device.
CGM Metric Time Below Range | 6 months
  Measures the percentage of time a participant's blood glucose levels fall below the target range using CGM device.
Summary of Diabetes Self Care Activities (SDSCA) Survey | 6 months
  Summary of Diabetes Self Care Activities Survey measures frequency and consistency of diabetes self-care activities during the past 7 days. Possible scores range from 0 (0 Days to 7 (7 Days). Higher scores indicate better compliance with diabetes self-care.
Diabetes Distress Scale | 6 months
  The Diabetes Distress Scale measures four critical dimensions of diabetes distress for participants: emotional, burden, regimen distress, interpersonal distress and physical distress. Possible scores range from 1 (Not a Problem) to 6 (A Very Serious Problem) with higher scores indicating higher levels of diabetes-related distress.

CONTACTS AND LOCATIONS:
Overall Officials: Athena Philis-Tsimikas, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Whittier Diabetes Institute, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No